CLINICAL TRIAL: NCT02889198
Title: Evaluation of Go NAP SACC: A Pilot Study Evaluating the Nutrition Tool of the Web-based Tool Based on the NAP SACC Program
Brief Title: A Pilot Study Evaluating Go NAP SACC's Web-based Nutrition Tool for Child Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 14-0931
Record Dates: First submitted 2016-08-26; First posted 2016-09-05 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Environment Related Disease
Keywords: web-based tool; child, preschool; nutrition; implementation; child care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Centers in this group will be granted immediate access to the Go NAP SACC website following randomization with minimal support from a local technical assistance provider. The center director will have 4 months to use Go NAPSACC tools.
  Interventions: Behavioral: Go NAP SACC
- Control group (No Intervention): During the study, centers in this group will receive no intervention. However, they will be granted delayed access to the Go NAP SACC website and technical assistance support after post-intervention measures are collected.

INTERVENTIONS:
Behavioral: Go NAP SACC — Go NAP SACC is a suite of online tools designed to help child care programs improve their nutrition environment. Tools include: self-assessment, goal setting, action planning, and tips and materials. In addition to these online tools, local technical assistance providers offer center directors an orientation on how to use Go NAP SACC and minimal ongoing technical assistance.
  Arms: Intervention group

SUMMARY:
The purpose of this project is to evaluate the effectiveness of Go NAP SACC (Get online with Nutrition and Physical Activity Self-Assessment for Child Care), a suite of web-based tools designed to help child care programs improve their nutrition environment (specifically classrooms serving 3-5 year olds) over the course of 4 months.

DETAILED DESCRIPTION:
National data show that many children, even as young as 2-5 years old, have adopted unhealthy eating patterns and are overweight/obese. Interventions targeting early childhood are critical for reversing these trends. More than half of 3-6 year olds in the US are enrolled in center-based child care programs, where they spend more than 25 hours per week. For these children, the center's nutrition environment can influence developing preferences and habits and thereby, weight status. The Nutrition and Physical Activity Self-Assessment for Child Care (NAP SACC) was developed in 2002 to help child care providers improve their food and physical activity environments. Evaluations of NAP SACC have shown it to be efficacious, but the program's reliance on trained technical assistance professionals and in-person delivery limits its potential for large-scale dissemination, especially in low-resourced rural areas. Go NAP SACC was developed to overcome this challenge by providing tailored web-based tools and resources that allow child care providers to complete more of the program on their own. This study will evaluate Go NAP SACC to determine if web-based delivery can broaden dissemination of the program, particularly in low-resourced rural areas.

This project will use a randomized controlled design to evaluate the impact of Go NAP SACC on centers' nutrition environments. A sample of 40 child care centers will be recruited to take part. Participating centers will be randomized (1:1) into one of two arms: immediate access (intervention) or delayed access (control). Measures will be collected at two time points, baseline and post-intervention (4 months later), to assess change in centers' nutrition environment scores.

The sample of 40 licensed centers will be recruited from rural counties in North Carolina. To facilitate recruitment, county-level Smart Start partnerships (local organizations that have existing relationships with child care programs) will be asked to share information about the study with their local centers and compile a list of those who might be interested in participating. Then, trained research assistants will follow-up with interested centers by telephone to confirm interest and eligibility. To be eligible, a center must serve 3-5 year old children and have 2 preschool teachers willing to take part in measures along with the center director, have a quality rating of 2-5 stars (or be exempt from ratings), and not have participated in NAP SACC in the last 6 months. Centers directors will complete a memorandum of understanding and informed consent; and teachers will be given informational fact sheets (but will not be asked to sign consent).

Centers will be randomized following their completion of baseline measures. Those randomized into the intervention arm will be given immediate access to Go NAP SACC online tools. To facilitate their use, technical assistance providers from the local Smart Start partnerships will provide an in-person orientation to each center director to help them register, learn to navigate the website, and review a timeline for implementation. Center directors will then have 4 months to complete the self-assessment, select goals to work on, create action plans, and implement those plans using resources from the tips and materials library. Technical assistance staff will provide brief monthly check-ins (by telephone or email) to prompt continued efforts. Centers randomized into the control group will receive the same access and support just 4-6 months later (once post-intervention measures are complete).

To evaluate the impact of Go NAP SACC, centers' nutrition environments will be assessed at two timepoints: baseline and post-intervention. These assessments will use the self-report version of the Environment and Policy Assessment and Observation (EPAO-SR), which uses self-administered surveys completed by directors and preschool teachers. The EPAO-SR will be modified to focus solely on the nutrition environment (eliminating physical activity and screen time items).

The statistical analysis will compare the differences in mean change in centers' nutrition environment scores from pre- to post-intervention between intervention and control groups. The analysis will assess change in the overall nutrition environment score, as well as changes in each of the seven environmental sub-components. Analyses will involve testing of the hypotheses under the intent-to-treat (ITT) principle using SAS v.9.2 and Generalized Linear Modeling (PROC GLM). Use of PROC GLM, instead of a simple t-test, will allow us to control for key characteristics (e.g., technical assistance staff, quality star rating, participation in Child and Adult Care Food Program). To further explore the effect of the intervention, the investigators will fit Generalized Linear Mixed Models that: 1) adjust for baseline variables distributed differently between the intervention and comparison groups; 2) test interaction terms between the treatment group and other covariates; and 3) examine completers only.

NOTE DEVIATION: While the anticipated sample was 40 child care centers, only 33 enrolled, 31 of which provided sufficient baseline and follow-up data to be included in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Child Care Centers must have a quality rating of 2-5 stars OR be licensed as GS110-106 (faith-based and exempt from rating), serve lunch and a snack, and have 3-4 year old classrooms and 2 preschool teacher willing to participate.
* Teachers must teach in the 3-4 year old classrooms.
* Center directors and teachers must be able to read English.

Exclusion Criteria:

* Child Care Centers cannot have participated in NAP SACC within the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in EPAO-SR Scores from Baseline to Post-intervention | Measures collected at baseline (2-4 weeks prior to the intervention) and post-intervention (1-3 weeks following the intervention)
  Nutrition-related environmental characteristics will be assessed using the EPAO-SR, integrating data from the center director, child care teachers, and trained staff (reviewing policy documents).Data from all components is used in scoring. Item responses are used to derive variables assessing compliance with 42 nutrition best practices (BPs). Each nutrition BP variable is scored on a 4-point scale (0-3), where higher scores indicate closer BP compliance. Nutrition BP variables are then sorted into one of 7 environmental components: foods provided (12), beverages provided (5), feeding practices (8), feeding environment (8), menus (1), education & professional development (6), or policy (1). Environmental summary scores are calculated by averaging scores from relevant nutrition BP variables; hence, summary scores range from 0 to 3. An overall nutrition score is calculated by summing the 7 environmental summary scores; hence overall nutrition scores range from 0 to 21.

CONTACTS AND LOCATIONS:
Overall Officials: Dianne S Ward, EdD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ward DS, Vaughn AE, Mazzucca S, Burney R. Translating a child care based intervention for online delivery: development and randomized pilot study of Go NAPSACC. BMC Public Health. 2017 Nov 21;17(1):891. doi: 10.1186/s12889-017-4898-z. PMID 29162057